CLINICAL TRIAL: NCT03870386
Title: EUS-guided Biliary Drainage of First Intent With the Lumen Apposing Metal Stent vs. ERCP in the Management of Malignant Distal Biliary Obstruction: a Randomized Controlled Trial
Brief Title: EUS Biliary Drainage vs. ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Yen-I Chen, Primary Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: F11-36171
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Biliary Obstruction
Keywords: EUS; ERCP; Lumen apposing metal stent; Biliary drainage; Biliary obstruction; Pancreatic adenocarcinoma
MeSH Terms: interventions — laminin beta2; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-BD with LAMS (Experimental): A curvilinear endoscope is inserted orally and advanced to the duodenal bulb. Biliary accessibility is confirmed via EUS and with Doppler to rule out any intervening vessels. For common bile ducts < 15 mm in diameter, the biliary access is established via needle puncture with a 19-gauge needle followed by advancement of a 0.035 or 0.025 inch guidewire. A LAMS (AxiosTM) will then be inserted with cautery assistance without tract dilation and deployed. For common bile ducts > 15 mm, the need for initial needle puncture and wire insertion is at the discretion of the endoscopist. A cholangiogram is then performed through the LAMS with contrast injection. The choice of stent size will be at the discretion of the endoscopist (8 x 8 mm or 6 x 8 mm).
  Interventions: Procedure: EUS-BD with LAMS
- Traditional transpapillary metal stent via ERCP (Active Comparator): A duodenoscope is advanced orally to the papilla. The bile duct is then cannulated with a sphincterotome using the guidewire-assisted technique. A cholangiogram is then performed followed by insertion of a self-expanding metal biliary stent. The performance of a biliary sphincterotomy prior to stent insertion and the choice of stent size (10x 40 mm, 10 x 60 mm, 10x 80 mm) will be at the discretion of the endoscopist.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: EUS-BD with LAMS — Endoscopic ultrasound guided insertion of lumen apposing metal stent forming a choledochoduodenostomy
  Arms: EUS-BD with LAMS
Procedure: ERCP — Endoscopic retrograde cholangiopancreatography to localize and cannulate the bile duct using the guidewire-assisted technique.
  Arms: Traditional transpapillary metal stent via ERCP

SUMMARY:
Endoscopic ultrasound guided biliary drainage (EUS-BD) is an evolving field that has grown in popularity in the management of malignant biliary obstruction. Although Endoscopic retrograde cholangio-pancreatography (ERCP) with stent insertion has been the mainstay therapy throughout several decades, the transpapillary approach through tumor tissue is associated with significant risk for adverse events such as post-ERCP pancreatitis and stent dysfunction from tumor tissue overgrowth and ingrowth. EUS-BD, through the creation of a choledochoduodenostomy with a stent, has the potential advantage of avoiding the papilla and its associated complications while potentially improving stent patency with lower risks for tumor tissue ingrowth and/or overgrowth.

ELIGIBILITY:
Inclusion Criteria:

* Radiological diagnosis (with or without pathological diagnosis) of borderline resectable, locally advanced, or unresectable malignant distal biliary obstruction at least 2 cm distal to the hilum. Resectability based on tumor staging on axial imaging and surgeon evaluation.
* Elevated liver tests with serum bilirubin at least 3 times above the upper limit of normal (18.9 umol/L)
* Dilated extra-hepatic bile duct measuring at least 1.2 cm on axial imaging or US
* Confirmation of bile duct accessibility and size of at least 1.2 cm on endoscopic ultrasound
* Karnofsky index > 30%
* ASA score <IV
* Provision of informed consent

Exclusion Criteria:

* Hilar obstruction (biliary obstruction < 2 cm from the hilum)
* Uncorrectable coagulopathy and/or thrombocytopenia
* Age < 18
* Liver metastasis involving > 30% of the liver volume
* Liver cirrhosis with portal hypertension or ascites
* Prior biliary sphincterotomy or stent placement
* Surgically altered anatomy
* Common bile duct measuring less than 1.2 cm will be excluded
* Patient with clinical and radiological evidence of gastric outlet obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of re-intervention | 1 year
  Obstruction and/or migration of stent

SECONDARY OUTCOMES:
Technical success | 1 year
  successful insertion of a transpapillary stent or choledochoduodenostomy stent at the initial procedure at time of randomization
Clinical success | 1 year
  50% decrease in bilirubin < 2 weeks post-stent insertion or less than 25% of pre-procedure bilirubin level within 4 weeks post stent insertion
Stent patency | 1 year
  mean time to stent obstruction or migration
Early adverse events | 1 year
  as per the ASGE lexicon for endoscopic adverse events13 including post-procedural pancreatitis defined as new or worsening abdominal pain persistent for at least 24 hours and requiring analgesics after ERCP or EUS-BD with an elevated amylase or lipase of greater than three times the upper limit of normal, peri-procedural bleeding defined as hematemesis and/or melena or hemoglobin drop > 2 g, intestinal perforation defined as evidence of air or luminal contents outside the GI tract, and cholangitis >38 Celsius for greater than 24 hours with cholestatic liver enzymes

CONTACTS AND LOCATIONS:
Overall Officials: Yen-I Chen, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (11):
- Canada (10):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, Bristish Columbia
  - St-Paul Hospital, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - St-Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier Universite de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hopital Charles Lemoynes, Montreal, Quebec
  - Jewish General Hospital, Montreal
- Hôpital Privé des Peupliers, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boulay BR, Lo SK. Endoscopic Ultrasound-Guided Biliary Drainage. Gastrointest Endosc Clin N Am. 2018 Apr;28(2):171-185. doi: 10.1016/j.giec.2017.11.005. Epub 2018 Feb 3. PMID 29519330
- [Background] Khashab MA, Messallam AA, Penas I, Nakai Y, Modayil RJ, De la Serna C, Hara K, El Zein M, Stavropoulos SN, Perez-Miranda M, Kumbhari V, Ngamruengphong S, Dhir VK, Park DH. International multicenter comparative trial of transluminal EUS-guided biliary drainage via hepatogastrostomy vs. choledochoduodenostomy approaches. Endosc Int Open. 2016 Feb;4(2):E175-81. doi: 10.1055/s-0041-109083. Epub 2016 Jan 15. PMID 26878045
- [Background] Khashab MA, Van der Merwe S, Kunda R, El Zein MH, Teoh AY, Marson FP, Fabbri C, Tarantino I, Varadarajulu S, Modayil RJ, Stavropoulos SN, Penas I, Ngamruengphong S, Kumbhari V, Romagnuolo J, Shah R, Kalloo AN, Perez-Miranda M, Artifon EL. Prospective international multicenter study on endoscopic ultrasound-guided biliary drainage for patients with malignant distal biliary obstruction after failed endoscopic retrograde cholangiopancreatography. Endosc Int Open. 2016 Apr;4(4):E487-96. doi: 10.1055/s-0042-102648. Epub 2016 Mar 30. PMID 27092334
- [Background] Almadi MA, Barkun A, Martel M. Plastic vs. Self-Expandable Metal Stents for Palliation in Malignant Biliary Obstruction: A Series of Meta-Analyses. Am J Gastroenterol. 2017 Feb;112(2):260-273. doi: 10.1038/ajg.2016.512. Epub 2016 Nov 15. PMID 27845340
- [Background] Almadi MA, Barkun JS, Barkun AN. Stenting in Malignant Biliary Obstruction. Gastrointest Endosc Clin N Am. 2015 Oct;25(4):691-711. doi: 10.1016/j.giec.2015.06.002. Epub 2015 Aug 28. PMID 26431598
- [Background] American Society for Gastrointestinal Endoscopy (ASGE) Standards of Practice Committee; Anderson MA, Appalaneni V, Ben-Menachem T, Decker GA, Early DS, Evans JA, Fanelli RD, Fisher DA, Fisher LR, Fukami N, Hwang JH, Ikenberry SO, Jain R, Jue TL, Khan K, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Shergill AK, Dominitz JA, Cash BD. The role of endoscopy in the evaluation and treatment of patients with biliary neoplasia. Gastrointest Endosc. 2013 Feb;77(2):167-74. doi: 10.1016/j.gie.2012.09.029. Epub 2012 Dec 7. No abstract available. PMID 23219047
- [Background] Bang JY, Navaneethan U, Hasan M, Hawes R, Varadarajulu S. Stent placement by EUS or ERCP for primary biliary decompression in pancreatic cancer: a randomized trial (with videos). Gastrointest Endosc. 2018 Jul;88(1):9-17. doi: 10.1016/j.gie.2018.03.012. Epub 2018 Mar 21. PMID 29574126
- [Background] Lee TH, Choi JH, Park do H, Song TJ, Kim DU, Paik WH, Hwangbo Y, Lee SS, Seo DW, Lee SK, Kim MH. Similar Efficacies of Endoscopic Ultrasound-guided Transmural and Percutaneous Drainage for Malignant Distal Biliary Obstruction. Clin Gastroenterol Hepatol. 2016 Jul;14(7):1011-1019.e3. doi: 10.1016/j.cgh.2015.12.032. Epub 2015 Dec 31. PMID 26748220
- [Background] Paik WH, Lee TH, Park DH, Choi JH, Kim SO, Jang S, Kim DU, Shim JH, Song TJ, Lee SS, Seo DW, Lee SK, Kim MH. EUS-Guided Biliary Drainage Versus ERCP for the Primary Palliation of Malignant Biliary Obstruction: A Multicenter Randomized Clinical Trial. Am J Gastroenterol. 2018 Jul;113(7):987-997. doi: 10.1038/s41395-018-0122-8. Epub 2018 Jul 2. PMID 29961772
- [Background] Park JK, Woo YS, Noh DH, Yang JI, Bae SY, Yun HS, Lee JK, Lee KT, Lee KH. Efficacy of EUS-guided and ERCP-guided biliary drainage for malignant biliary obstruction: prospective randomized controlled study. Gastrointest Endosc. 2018 Aug;88(2):277-282. doi: 10.1016/j.gie.2018.03.015. Epub 2018 Mar 30. PMID 29605722
- [Background] Kunda R, Perez-Miranda M, Will U, Ullrich S, Brenke D, Dollhopf M, Meier M, Larghi A. EUS-guided choledochoduodenostomy for malignant distal biliary obstruction using a lumen-apposing fully covered metal stent after failed ERCP. Surg Endosc. 2016 Nov;30(11):5002-5008. doi: 10.1007/s00464-016-4845-6. Epub 2016 Mar 11. PMID 26969661
- [Background] Anderloni A, Fugazza A, Troncone E, Auriemma F, Carrara S, Semeraro R, Maselli R, Di Leo M, D'Amico F, Sethi A, Repici A. Single-stage EUS-guided choledochoduodenostomy using a lumen-apposing metal stent for malignant distal biliary obstruction. Gastrointest Endosc. 2019 Jan;89(1):69-76. doi: 10.1016/j.gie.2018.08.047. Epub 2018 Sep 4. PMID 30189198
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Liao WC, Chien KL, Lin YL, Wu MS, Lin JT, Wang HP, Tu YK. Adjuvant treatments for resected pancreatic adenocarcinoma: a systematic review and network meta-analysis. Lancet Oncol. 2013 Oct;14(11):1095-1103. doi: 10.1016/S1470-2045(13)70388-7. Epub 2013 Sep 12. PMID 24035532
- [Background] Freeman ML, Nelson DB, Sherman S, Haber GB, Herman ME, Dorsher PJ, Moore JP, Fennerty MB, Ryan ME, Shaw MJ, Lande JD, Pheley AM. Complications of endoscopic biliary sphincterotomy. N Engl J Med. 1996 Sep 26;335(13):909-18. doi: 10.1056/NEJM199609263351301. PMID 8782497
- [Background] Kochar B, Akshintala VS, Afghani E, Elmunzer BJ, Kim KJ, Lennon AM, Khashab MA, Kalloo AN, Singh VK. Incidence, severity, and mortality of post-ERCP pancreatitis: a systematic review by using randomized, controlled trials. Gastrointest Endosc. 2015 Jan;81(1):143-149.e9. doi: 10.1016/j.gie.2014.06.045. Epub 2014 Aug 1. PMID 25088919
- [Background] Almadi MA, Barkun A, Martel M. Self-expandable metal stents versus plastic stents for malignant biliary obstruction. Gastrointest Endosc. 2016 Apr;83(4):852-3. doi: 10.1016/j.gie.2015.10.035. No abstract available. PMID 26975289
- [Background] Gardner TB, Spangler CC, Byanova KL, Ripple GH, Rockacy MJ, Levenick JM, Smith KD, Colacchio TA, Barth RJ, Zaki BI, Tsapakos MJ, Gordon SR. Cost-effectiveness and clinical efficacy of biliary stents in patients undergoing neoadjuvant therapy for pancreatic adenocarcinoma in a randomized controlled trial. Gastrointest Endosc. 2016 Sep;84(3):460-6. doi: 10.1016/j.gie.2016.02.047. Epub 2016 Mar 10. PMID 26972022
- [Background] Barkun AN, Adam V, Martel M, AlNaamani K, Moses PL. Partially covered self-expandable metal stents versus polyethylene stents for malignant biliary obstruction: a cost-effectiveness analysis. Can J Gastroenterol Hepatol. 2015 Oct;29(7):377-83. doi: 10.1155/2015/743417. Epub 2015 Jun 30. PMID 26125107
- [Background] Yachimski PS, Ross A. The Future of Endoscopic Retrograde Cholangiopancreatography. Gastroenterology. 2017 Aug;153(2):338-344. doi: 10.1053/j.gastro.2017.06.015. Epub 2017 Jun 21. No abstract available. PMID 28647354
- [Background] Giovannini M, Moutardier V, Pesenti C, Bories E, Lelong B, Delpero JR. Endoscopic ultrasound-guided bilioduodenal anastomosis: a new technique for biliary drainage. Endoscopy. 2001 Oct;33(10):898-900. doi: 10.1055/s-2001-17324. PMID 11571690
- [Background] Sharaiha RZ, Khan MA, Kamal F, Tyberg A, Tombazzi CR, Ali B, Tombazzi C, Kahaleh M. Efficacy and safety of EUS-guided biliary drainage in comparison with percutaneous biliary drainage when ERCP fails: a systematic review and meta-analysis. Gastrointest Endosc. 2017 May;85(5):904-914. doi: 10.1016/j.gie.2016.12.023. Epub 2017 Jan 4. PMID 28063840
- [Background] Binmoeller KF, Shah JN. Endoscopic ultrasound-guided gastroenterostomy using novel tools designed for transluminal therapy: a porcine study. Endoscopy. 2012 May;44(5):499-503. doi: 10.1055/s-0032-1309382. Epub 2012 Apr 24. PMID 22531985
- [Background] Chen YI, Kunda R, Storm AC, Aridi HD, Thompson CC, Nieto J, James T, Irani S, Bukhari M, Gutierrez OB, Agarwal A, Fayad L, Moran R, Alammar N, Sanaei O, Canto MI, Singh VK, Baron TH, Khashab MA. EUS-guided gastroenterostomy: a multicenter study comparing the direct and balloon-assisted techniques. Gastrointest Endosc. 2018 May;87(5):1215-1221. doi: 10.1016/j.gie.2017.07.030. Epub 2017 Jul 24. PMID 28750837
- [Background] Kamarajah SK, Burns WR, Frankel TL, Cho CS, Nathan H. Validation of the American Joint Commission on Cancer (AJCC) 8th Edition Staging System for Patients with Pancreatic Adenocarcinoma: A Surveillance, Epidemiology and End Results (SEER) Analysis. Ann Surg Oncol. 2017 Jul;24(7):2023-2030. doi: 10.1245/s10434-017-5810-x. Epub 2017 Feb 17. PMID 28213792
- [Derived] Chen YI, Sahai A, Donatelli G, Lam E, Forbes N, Mosko J, Paquin SC, Donnellan F, Chatterjee A, Telford J, Miller C, Desilets E, Sandha G, Kenshil S, Mohamed R, May G, Gan I, Barkun J, Calo N, Nawawi A, Friedman G, Cohen A, Maniere T, Chaudhury P, Metrakos P, Zogopoulos G, Bessissow A, Khalil JA, Baffis V, Waschke K, Parent J, Soulellis C, Khashab M, Kunda R, Geraci O, Martel M, Schwartzman K, Fiore JF Jr, Rahme E, Barkun A. Endoscopic Ultrasound-Guided Biliary Drainage of First Intent With a Lumen-Apposing Metal Stent vs Endoscopic Retrograde Cholangiopancreatography in Malignant Distal Biliary Obstruction: A Multicenter Randomized Controlled Study (ELEMENT Trial). Gastroenterology. 2023 Nov;165(5):1249-1261.e5. doi: 10.1053/j.gastro.2023.07.024. Epub 2023 Aug 6. PMID 37549753
- [Derived] Chen YI, Callichurn K, Chatterjee A, Desilets E, Fergal D, Forbes N, Gan I, Kenshil S, Khashab MA, Kunda R, Lam E, May G, Mohamed R, Mosko J, Paquin SC, Sahai A, Sandha G, Teshima C, Barkun A, Barkun J, Bessissow A, Candido K, Martel M, Miller C, Waschke K, Zogopoulos G, Wong C; ELEMENT trial and for the Canadian Endoscopic Research Collaborative (CERC). ELEMENT TRIAL: study protocol for a randomized controlled trial on endoscopic ultrasound-guided biliary drainage of first intent with a lumen-apposing metal stent vs. endoscopic retrograde cholangio-pancreatography in the management of malignant distal biliary obstruction. Trials. 2019 Dec 9;20(1):696. doi: 10.1186/s13063-019-3918-y. PMID 31818329